CLINICAL TRIAL: NCT00799565
Title: Genetic Polymorphisms in Idiopathic Mitral Valve Prolapse :A French Prospective Study Using a Genome Wide Analysis
Brief Title: Mitral Valve Prolapse (MVP) - France Study
Acronym: MVP-France
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: French Cardiology Society (Other)
Collaborators: Leducq Foundation (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Centre National de Génotypage (Other)
Responsible Party: Pr Geneviève Derumeaux, French Society of Cardiology
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2008-01
Record Dates: First submitted 2008-11-24; First posted 2008-12-01 (Estimated); Last update posted 2011-07-14 (Estimated); Status verified 2011-07

CONDITIONS: Mitral Valve Prolapse
Keywords: Mitral Valve prolapse; echography; genetic study; study case-witness; Patients with a Mitral Valve Prolapse
MeSH Terms: conditions — Mitral Valve Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Subject with a Mitral Valvular Prolapse
  Interventions: Genetic: catch of blood
- 2 (Experimental): Healthy Volunteers
  Interventions: Genetic: catch of blood

INTERVENTIONS:
Genetic: catch of blood — 4 tubes of blood are taken on subjects. Samples are sent in Pr Jeunemaître to extract DNA and stock it.
  This DNA bank aims to search for susceptibility genes in MVP using a genome wide analysis and comparing results obtained in 1000 patients with MVP and 1000 non-MVP subjects

SUMMARY:
This prospective nation-wide (France) study aims to search for susceptibility genes in MVP using a genome wide analysis and comparing results obtained in 1000 patients with MVP and 1000 non-MVP subjects.

DETAILED DESCRIPTION:
Two MVP populations will be defined in that study, either with the classical Barlow (myxomatous) disease or the fibroelastic degenerescence (thin and redundant leaflets).

MVP adult patients (> 18 year-old) will be included if they present the following 1) or 2) criteria :

1. 2D-echocardiographic mitral leaflet prolapse on the parasternal long-axis view > 2 mm AND leaflet thickness > 4 mm or mitral regurgitation > 2 + (using color Doppler)
2. Previous surgery for pure severe mitral regurgitation due to MVP with Barlow disease or fibroelastic degenerescence (with operative report available)

Patients will be excluded in case of associated heart disease (hypertrophic cardiomyopathy, rheumatismal disease…) or syndromic disease (Marfan, Ehlers-Danlos…).

Around 30 (cardiology, cardiovascular surgery) french centers will participate to this study. An e-CRF will be used to collect clinical data. A genetic core lab will collect the DNA samples. An echocardiographic core lab will collect and read all the echo recordings.

DNA analysis will be compared between the patient group and spouses of the patients used as controls. In case of inadequacies concerning group size or age, available genotyped cohorts will be used.

ELIGIBILITY:
Inclusion criteria for MVP patients :

* Male or female subject ≥18 years
* Affiliation to the French social insurance system
* Written informed consent
* Idiopathic MVP defined by the presence of criteria 1) and 2) OR of criterion 3) :

  1. Echographic MVP > 2 mm on the left ventricular parasternal long-axis view
  2. Echographic myxomatous valve (thickness > 4 mm) or significant mitral regurgitation (> 2 + using color Doppler)
  3. History of mitral valve surgery for pure mitral regurgitation due to MVP (myxomatous or fibroelastic deficiency) with available detailed operative report.

Exclusion criteria :

* Presence of heart disease causing MVP (rheumatic, HCM…)
* Syndromic disease (Marfan, Ehlers-Danlos…)

Inclusion criteria for healthy subject :

* Male or female subject ≥40 years
* Absence of MVP or absence of mitral valve dystrophy
* Caucasian

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1179 (Actual)
Dates: Start 2008-12; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Genetic polymorphism identification | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Albert Alain Hagège, MD, PhD, Principal Investigator — Hôpital Européen Georges-Pompidou
Locations (26):
- France (26):
  - Hôpital Sud, Amiens
  - Clinique Saint Augustin, Bordeaux
  - Hôpital Ambroise Paré, Boulogne
  - Hôpital de la Cavale Blanche, Brest
  - Hôpital Gabriel Montpied, Clermont-Ferrand
  - Hôpital Henri Mondor, Créteil
  - Hôpital du Bocage, Dijon
  - Hôpital Front-Pré, La Seyne-sur-Mer
  - Hôpital Cardiologique, Lille
  - Hôpital Dupuytren, Limoges
  - Groupement Hospitalier Est, Lyon
  - Hôpital de la Timone, Marseille
  - Institut Hospitalier Jacques Cartier, Massy
  - Hôpital Arnaud de Villeneuve, Montpellier
  - Hôpital G and R Laennec, Nantes
  - Hôpital Lariboisière, Paris
  - Hôpital Pitié Salpêtrière, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Bichat, Paris
  - Hôpital Saint Antoine, Paris
  - Hôpital Cochin, Paris
  - Hôpital Cardiologique du Haut Lévêque, Pessac
  - Hôpital Pontchaillou, Rennes
  - Hôpital Charles Nicolle, Rouen
  - Hôpital Rangueil, Toulouse
  - CHU Nancy, Vandœuvre-lès-Nancy